CLINICAL TRIAL: NCT00503451
Title: A Phase IB, Study to Investigate the Effect of Ketoconazole, a CYP3A4 Inhibitor, on Oral LBH589 and to Assess the Efficacy and Safety of Oral LBH589 in Patients With Advanced Solid Tumors.
Brief Title: A Study to Investigate the Effects of Ketoconazole on LBH589 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2110
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-11

CONDITIONS: Non-Hodgkin Lymphoma; Neoplasms
Keywords: Advanced cancer; solid tumors; lymphoma; HDAC; LBH589; adults; non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms; Lymphoma | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589
  Other Names: Panobinostat

SUMMARY:
The primary purpose of this open-label study is to investigate the interaction of ketoconazole, a liver enzyme inhibitor, on oral LBH589 in adult patients with advanced solid tumors. The extension phase of the study will evaluate the safety and efficacy of LBH589 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically confirmed solid tumors or non-Hodgkin's lymphoma with progression on prior standard therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Adequate kidney function and laboratory values

Exclusion criteria:

* Patients who have received chemotherapy, any investigational drug, undergone major surgery, or received wide field radiotherapy less than 4 weeks ago
* Patients who had a heart attack or have unstable angina within past 6 months
* Heart disease including congestive heart failure and uncontrolled high blood pressure
* Liver disease, abnormal gastrointestinal (GI) function or ongoing diarrhea
* Use of any anti-cancer therapy, including radiation therapy, or certain drugs while on study
* Female patients who are pregnant or breast feeding.

Other protocol inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Levels of LBH589 in the blood on days 1, 5, 8, 9 and 10 of first cycle | 2 weeks

SECONDARY OUTCOMES:
Safety, tolerability and efficacy of oral LBH589 throughout the study | at least every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Nevada Cancer Institute, Las Vegas, Nevada, United States
- Novartis Investigative Site, Rotterdam, Netherlands

REFERENCES:
- [Derived] Hamberg P, Woo MM, Chen LC, Verweij J, Porro MG, Zhao L, Li W, van der Biessen D, Sharma S, Hengelage T, de Jonge M. Effect of ketoconazole-mediated CYP3A4 inhibition on clinical pharmacokinetics of panobinostat (LBH589), an orally active histone deacetylase inhibitor. Cancer Chemother Pharmacol. 2011 Sep;68(3):805-13. doi: 10.1007/s00280-011-1693-x. Epub 2011 Jun 26. PMID 21706316
- See also: Results for CLBH589B2110 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4102